CLINICAL TRIAL: NCT02991170
Title: Impact of Radiofrequency Ablation Therapy in Coronary Artery Bypass Grafts Surgery on Outcomes in Patients With Myocardial Infarction Related Ventricular Arrhythmia
Brief Title: Effect of Radiofrequency Ablation in Patients With Ventricular Arrhythmia Undergoing CABG
Acronym: RACAVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Yang Yu, Deputy Director of Cardiac Surgery, Principal Investigator,Clinical Professor, Beijing Anzhen Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XMLX201504
Record Dates: First submitted 2016-12-07; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: MI Related Malignant Ventricular Arrhythmia
Keywords: myocardial infarction; ventricular arrhythmia; radiofrequency ablation; Coronary Artery Bypass Grafts
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Active Comparator): Patients with myocardial infarction related potential malignant ventricular arrhythmia undergoing Coronary Artery Bypass Grafts
  Interventions: Procedure: CABG
- interventional group (Experimental): Patients with myocardial infarction related potential malignant ventricular arrhythmia undergoing unipolar or bipolar radiofrequency ablation and Coronary Artery Bypass Grafts at the same time
  Interventions: Procedure: unipolar or bipolar radiofrequency ablation+CABG

INTERVENTIONS:
Procedure: unipolar or bipolar radiofrequency ablation+CABG — Patients with myocardial infarction related potential malignant ventricular arrhythmia undergoing unipolar or bipolar radiofrequency ablation and Coronary Artery Bypass Grafts at the same time
  Arms: interventional group
Procedure: CABG — Patients with myocardial infarction related potential malignant ventricular arrhythmia undergoing Coronary Artery Bypass Grafts
  Arms: control group

SUMMARY:
Patients with myocardial infarction related potential malignant ventricular arrhythmia have high risk of sudden death. The aim of this clinical trial is evaluating therapeutic efficacy of unipolar or bipolar radiofrequency ablation in Coronary Artery Bypass Grafts (CABG) Surgery, which can reduce myocardial ischemia and block reentry circuits of ventricular arrhythmia at the same time. The observation indexes include the morbidity of potential malignant ventricular arrhythmia and major adverse cardiovascular events in mid-long-term after CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patients have been receiving coronary artery bypass grafts from 2015.1-2017.12
* The patients had old myocardial infarction related potential malignant ventricular arrhythmia
* Anti-arrhythmic drug treatment is invalid
* All enrolled patients must being signed the informed consent

Exclusion Criteria:

* Severe heart failure( ejection fraction under 35%)
* Patients with acute myocardial infarction
* Patients with ICD implanted

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Morbidity of potential malignant ventricular arrhythmia | 1 year after surgery
  The morbidity of potential malignant ventricular arrhythmia in 1 year after surgery

SECONDARY OUTCOMES:
Morbidity of major adverse cardiovascular events | 1 year after surgery
  The morbidity of the major adverse cardiovascular events in 1 year after surgery

OTHER OUTCOMES:
Cardiac function | Change from Baseline Cardiac Function at 3 month, 6 month, 1 year, 2 year after surgery
  Change from Baseline Cardiac Function evaluated by echocardiography at 3 month, 6 month, 1 year, 2 year after surgery
Cardiac electrophysiology index | Change from Baseline Cardiac Electrophysiology Index at 1 year and 2 year after surgery
  Change from Baseline Cardiac Electrophysiology Index evaluated by Holter and cardiac magnetic resonance imaging or CARTO at 1 year and 2 year after surgery
Seattle Angina Questionnaire | Change from Baseline Seattle Angina Questionnaire at 3 month, 6 month, 1 year, 2 year after surgery
  Change from Baseline the Seattle Angina Questionnaire at 3 month, 6 month, 1 year, 2 year after surgery

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Xuanwu Hospital, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided